CLINICAL TRIAL: NCT06239402
Title: Prospective Observational Study on the Therapeutic Strategy with Direct Oral Anticoagulants and Antiaggregant Drugs in Ischemic Heart Disease (PRODOAC)
Brief Title: Therapeutic Strategy with Direct Oral Anticoagulants and Antiaggregant Drugs in Ischemic Heart Disease
Acronym: PRODOAC
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Società Italiana Cardiologia Ospedalità Accreditata (SICOA) (Unknown)
Responsible Party: Principal Investigator, Laura Adelaide Dalla Vecchia, Principal Investigator, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: 2365CE
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observation — Observation of mortality, haemorrhagic and ischemic events in the studied population

SUMMARY:
The study aims to depict the actual prescription patterns employed in clinical practice of patients affected by non-valvular atrial fibrillation undergoing percutaneous coronary intervention (i.e. with a therapeutic indication for dual or triple antithrombotic therapy) and to analyze the outcomes of therapeutic decisions, focusing on mortality, hemorrhagic events, and ischemic events,

DETAILED DESCRIPTION:
The combination of warfarin, aspirin, and clopidogrel represented the standard antithrombotic therapeutic strategy for patients with atrial fibrillation and suffering from acute coronary syndrome and/or undergoing percutaneous coronary intervention.

Current guidelines and clinical practice guides suggest the use of triple or dual antithrombotic therapy after a careful evaluation of the patient's hemorrhagic and thrombotic profile, without however providing indications with recommendation class I. It is not known what treatment regimens are prescribed in the real world, i.e. how clinicians behave in the absence of clear guidelines.

This observational study involves patients affected by non-valvular atrial fibrillation undergoing percutaneous coronary intervention (i.e. with a therapeutic indication for dual or triple antithrombotic therapy), to describe the real-world prescription model used in clinical practice and to analyze the results of therapeutic choices in terms of mortality, hemorrhagic and ischemic events.

Patients are enrolled within 7 days from percutaneous coronary intervention during their hospitalization period. During the enrolment visit (i.e. baseline, T0), all patients undergo a detailed assessment of their medical history related to the recent hospitalization, laboratory blood analysis, and data related to their cardiovascular risk factors. Follow-up visits will be performed at three months (T3) and twelve months (T12). During the follow-up visit, any ischemic/bleeding events, therapeutic changes, and laboratory blood analysis will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non valvular atrial fibrillation with direct oral anticoagulants therapy
* Patient on antiplatelet therapy (acetylsalicylic acid and/or inhibitor of the P2Y12 platelet receptor)
* Patient hospitalized for percutaneous coronary intervention in the previous 7 days
* Age ≥18 years
* Estimated life expectancy ≥ 12 months
* Ability to give informed consent

Exclusion Criteria:

* Patients who have contraindications to direct oral anticoagulants therapy
* Patients who are indicated for direct oral anticoagulants therapy for reasons other than non valvular atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with non valvular atrial fibrillation with direct oral anticoagulants and antiplatelet therapy who underwent percutaneous coronary intervention in the previous 7 days
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Bleeding | 3 months
  Incidence of major bleeding and clinically relevant non major bleeding
Bleeding | 12 months
  Incidence of major bleeding and clinically relevant non major bleeding

SECONDARY OUTCOMES:
Adverse events | 3 months
  Cardiovascular events, death
Adverse events | 12 months
  Cardiovascular events, death

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri, Milan, Italy

IPD SHARING:
Plan to Share IPD: No